CLINICAL TRIAL: NCT05770596
Title: Impact of Perioperative Vitamin C on Acute and Chronic Post Mastectomy Pain After Breast Cancer Surgery
Brief Title: Vitamin C on Acute and Chronic Post Mastectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Rehab, Lecturer of anesthesiology, S.I.C.U and pain medicine Tanta university, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR116/2/23
Record Dates: First submitted 2023-03-05; First posted 2023-03-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Vitamin C; Post-mastectomy Pain Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C group (Experimental): patients in this group will receive 2 gm vitamin C orally 1 hour before surgery and will receive 0.5 gm vitamin C per day orally for 50 days starting from the 2nd postoperative day.
  Interventions: Drug: vitamin C group
- Placebo group (Placebo Comparator): patients in this group will receive placebo tablets with the same manner.1 hour before surgery and for 50 days starting from the 2nd postoperative day.
  Interventions: Other: placebo group

INTERVENTIONS:
Drug: vitamin C group — patients in this group will receive 2 gm vitamin C orally 1 hour before surgery and will receive 0.5 gm vitamin C per day orally for 50 days starting from the 2nd postoperative day.
  Arms: Vitamin C group
Other: placebo group — patients in this group will receive placebo tablets with the same manner; orally 1 hour before surgery and for 50 days starting from the 2nd postoperative day.
  Arms: Placebo group

SUMMARY:
This prospective randomized double-blinded controlled study will be conducted to evaluate the effect of perioperative vitamin C on acute and chronic post mastectomy pain after breast cancer surgery

DETAILED DESCRIPTION:
There is cumulative evidence that postoperative pain is closely associated with subsequent persistent pain lasting months. The International Association for the Study of Pain has defined chronic postsurgical pain (CPSP) as a pain that develops after surgical intervention and persists at least 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18years, with primary unilateral breast cancer and scheduled for lumpectomy, partial or total mastectomy with or without axillary lymph node dissection or modified radical mastectomy.

Exclusion Criteria:

- (1) Patients with renal stones or renal insufficiency, patients suffering from nausea and vomiting, gastroesophageal reflux or patients with chronic pain state.

(2) Intake of analgesic within 24 hours before surgery. (3) Patients unable to comply with the study protocol for any reason. (4) Contraindications to paravertebral block (PVB) such as allergy to local anesthetics, infection, or coagulopathy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients aged ≥ 18years, with primary unilateral breast cancer and scheduled for lumpectomy, partial or total mastectomy with or without axillary lymph node dissection or modified radical mastectomy.
Enrollment: 204 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
The incidence of chronic post mastectomy pain | 6 months after surgery
  Chronic pain will be assessed at 3, 6 months after surgery. Chronic pain will be defined as pain at the surgical site greater than or equal to 3 out of 10 on item 5 of the Brief Pain Inventory (item 5: "Please rate your pain by circling the one number that best describes your pain on the average in the past 24h, no pain = 0, worst pain = 10")

SECONDARY OUTCOMES:
The degree of acute postoperative pain | 48 hours postoperative
  degree of acute postoperative pain scores in the 1st and 2nd postoperative days using visual analogue scale (VAS) in both groups.
  Postoperative pain using VAS scores: will be assessed at 1, 4, 6, 12, 18, 24, 30, 36, 42 and 48 hr. after surgery.
  0: No pain, 10: the worst pain
The amount of total opioid dose in 48 hours after surgery | 48 hours postoperative
  Postoperative pain in the 1st and 2nd days will be assessed using VAS scores. If VAS score more than or equal to 4, morphine 0.05 mg/kg will be given.
The incidence of adverse effects | 48 hours postoperative
  postoperative adverse effects like postoperative nausea and vomiting (PONV).
The incidence of chronic pain at 9, 12 months after surgery | 12 months after surgery
  Chronic pain will be assessed at 9, 12 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be available upon a reasonable request from the corresponding author after the end of study for 1 year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.